CLINICAL TRIAL: NCT02287610
Title: A Non-Interventional Study to Evaluate the Effectiveness of Delayed-Release Prednisone (RAYOS) on Clinical Assessments and Serologic Disease Activity in Patients With Active Rheumatoid Arthritis in the Clinical Practice Setting
Brief Title: A Non-Interventional Study of RAYOS in Adult Patients With Rheumatoid Arthritis
Acronym: SUNRAY
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: HZ-PRE-NIS02
Record Dates: First submitted 2014-11-06; First posted 2014-11-10 (Estimated); Results first posted 2017-02-03 (Estimated); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Rheumatoid Arthritis
Keywords: RA; Delayed-release prednisone; Immediate-release prednisone; Non-interventional
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: RAYOS (delayed-release prednisone) — Physicians may prescribe any dosage of RAYOS based on what is appropriate for the treatment of the patient's condition as determined by performing standard of care assessments.

SUMMARY:
The overall objective of the study is to assess the effectiveness of switching from immediate-release prednisone (conventional) therapy to delayed-release prednisone (RAYOS) in patients with moderately to severely active Rheumatoid Arthritis (RA), managed according to standard of care in clinical practice settings.

DETAILED DESCRIPTION:
Adult Rheumatoid Arthritis (RA) participants previously receiving immediate release prednisone were enrolled in the trial if they and their physicians both consented. Once entered, participant baseline data were captured and they were switched to delayed-release prednisone and followed for approximately 12 weeks.

Study with completed results acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and in general good health (Investigator discretion) with a recent stable medical history other than related to RA disease activity
* RA diagnosis is ≥ 6 months according to ACR and/or EULAR classification criteria for diagnosis of active RA
* Morning stiffness duration of at least 45 minutes at study entry
* RA disease activity as defined by DAS28 of ≥ 3.2 at study entry
* Currently receiving conventional immediate-release prednisone ≥ 2.5 milligram (mg) every morning and previously agreed to switch to RAYOS
* Willing and able to sign an Informed Consent Form (ICF)

Exclusion Criteria:

* Patient is unwilling to participate in the non-interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult males and females with moderately to severely active disease who have previously received immediate-release prednisone (conventional) therapy, and prior to enrolling the SUNRAY Study, have made the joint decision (with their physicians) to convert to delayed-release prednisone (RAYOS).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Dikranian AH, Mallay R, Marshall M, Francis-Sedlak M, Holt RJ. Switching From Immediate-Release to Delayed-Release Prednisone in Moderate to Severe Rheumatoid Arthritis: A Practice-Based Clinical Study. Rheumatol Ther. 2017 Dec;4(2):363-374. doi: 10.1007/s40744-017-0075-1. Epub 2017 Aug 17. PMID 28819927

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total, 75 participants enrolled in the study, 11 of them did not meet eligibility requirements and therefore were not included.
Groups:
- Delayed-release Prednisone (RAYOS): Adult Rheumatoid Arthritis (RA) participants previously receiving immediate release prednisone were enrolled in the trial if they and their physicians both consented. Once entered, participant baseline data were captured and they were switched to delayed-release prednisone at the same dose of prednisone previously received.
Period: Overall Study
Arm/Group | Delayed-release Prednisone (RAYOS)
Started | 64
Per Protocol Follow-Up | 56
Completed | 48
Not Completed | 16
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 8
Not completed — Excluded-investigator non-responsiveness | 5

BASELINE CHARACTERISTICS:
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.05 (12.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 12
Age at Rheumatoid Arthritis Diagnosis [Mean (Standard Deviation); unit: years] | 56.49 (14.69)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Severity of Morning Stiffness (Using 100mm VAS) From Baseline (Week 0) to Final Follow-Up Visit
Description: Mean change in severity of morning stiffness was assessed using a 0 to 100 millimeter (mm) Visual Analogue Scale (VAS) where 0 corresponded to "Not Severe at All" and 100 to "Extremely Severe". This measure was collected at baseline and at the last follow-up visit. As this study was a non-interventional research initiative and no assessments or visits were mandated, the mean change was only calculated for participants that had measurements at both baseline and final follow-up.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: 56 participants were in the per protocol follow-up analysis set. Mean change in severity of morning stiffness was calculated for participants who had both baseline and follow-up severity of morning stiffness data. For severity of morning stiffness, the mean change from baseline is based on 38 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 38
units on a scale | -5.2 (27.3)

2. Secondary Outcome: Change in Duration of Morning Stiffness (Minutes) From Baseline to Final Visit (Final Follow-Up Visit)
Description: The duration of morning stiffness was the amount of time participants experienced stiffness after getting up in the morning. This measure was collected at baseline and at the last follow-up visit. As this study was a non-interventional research initiative and no assessments or visits were mandated, the change in duration of morning stiffness was only calculated for participants that had measurements at both baseline and final follow-up.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: 56 participants were in the per protocol follow-up analysis set. The change in duration of morning stiffness (minutes) was calculated for participants who had both baseline and follow-up morning stiffness data. For duration of morning stiffness, the mean change from baseline is based on 41 participants.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 41
minutes | -18.9 (77.5)

3. Secondary Outcome: Change in Patient's Overall Assessment in Disease Activity From Baseline to Final Visit (Final Follow-up Visit)
Description: Patient's Overall Assessment in Disease Activity was measured by asking the participant to rate on a 10-cm visual analogue scale (VAS) how well they were doing considering all of the ways their arthritis affected them: 0 - Very Well, 10 - Very Poor. As this study was a non-interventional research initiative and no assessments or visits were mandated, the change in Patient's Overall Assessment in Disease Activity was only calculated for participants that had measurements at both baseline and final follow-up.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: 56 participants were in the per protocol follow-up analysis set. Change in Patient's Overall Assessment in Disease Activity was calculated for participants who had both baseline and follow-up Patient's Overall Assessment in Disease Activity data. For this measure, the mean change from baseline is based on 36 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 36
units on a scale | -0.47 (2.40)

4. Secondary Outcome: Change in Physician's Overall Assessment in Disease Activity From Baseline to Final Visit (Final Follow-up Visit)
Description: Physician's Overall Assessment in Disease Activity was measured with a 10-cm visual analogue scale (VAS) where 0 corresponded to "Very Well' and 10 to "Very Poor". As this study was a non-interventional research initiative and no assessments or visits were mandated, the change in Physician's Overall Assessment in Disease Activity was only calculated for participants that had measurements at both baseline and final follow-up.
Time Frame: Baseline to Last Follow-up visit (up to 18.7 weeks)
Population: 56 participants were in the per protocol follow-up analysis set. Change in Physician's Overall Assessment in Disease Activity was calculated for participants who had both baseline and follow-up Physician's Overall Assessment in Disease Activity data. For this measure, the mean change from baseline is based on 37 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 37
units on a scale | -0.86 (2.34)

5. Secondary Outcome: Change in Disease Activity Score in 28 Joints Calculated With Erythrocyte Sedimentation Rate (DAS28-ESR) From Baseline to Final Visit (Final Follow-up Visit)
Description: The DAS28 is an index for measuring disease activity in rheumatoid arthritis (RA). The index includes swollen joint counts (SJC) and tender joint counts (TJC), both scored 0-28 (higher scores indicate higher disease activity), as well as acute phase response determined by erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP), and patient global assessment (PGA) on a visual analogue scale (higher scores indicate higher disease activity).
  DAS28-ESR was calculated according to the following formula: DAS28-ESR equals (=) [0.56 multiplied by (*) the square root (√) of TJC] plus (+) [0.28 * √ of SJC] + [0.70 * the natural logarithm (ln) ESR in millimeters per hour (mm/h)] + [0.014 * PGA in mm]. A negative change from baseline indicates improvement.
  As this study was a non-interventional research initiative and no assessments or visits were mandated, the change in DAS28-ESR was only calculated for participants that had measurements at both baseline and final follow-up.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: 56 participants were in the per protocol follow-up analysis set. Change in DAS28-ESR was calculated for participants who had both baseline and follow-up data required to calculate DAS28-ESR. For this measure, the mean change from baseline is based on 15 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 15
units on a scale | -0.39 (1.10)

6. Secondary Outcome: Change in Disease Activity Score in 28 Joints Calculated With C-reactive Protein (DAS28-CRP) From Baseline to Final Visit (Final Follow-up Visit)
Description: The DAS28 is an index for measuring disease activity in rheumatoid arthritis (RA). The index includes swollen joint counts (SJC) and tender joint counts (TJC), both scored 0-28 (higher scores indicate higher disease activity), as well as acute phase response determined by erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP), and patient global assessment (PGA) on a visual analogue scale (higher scores indicate higher disease activity).
  DAS28-CRP was calculated according to the following formula: DAS28-CRP equals (=) [0.56 multiplied by (*) the square root (√) of TJC] plus (+) [0.28 * √ of SJC] + [0.36 * the natural logarithm (ln) of (CRP + 1)] + [0.014 * PGA in mm] + 0.96. A negative change from baseline indicated improvement.
  As this study was a non-interventional research initiative and no assessments or visits were mandated, the change in DAS28-CRP was only calculated for participants that had measurements at both baseline and final follow-up.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: 56 participants were in the per protocol follow-up analysis set. Change in Disease Activity Score in 28 Joints calculated with C-reactive protein (DAS28-CRP) was calculated for participants who had both baseline and follow-up data required to calculate DAS28-CRP. For this measure, the mean change from baseline is based on 25 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 25
units on a scale | -0.62 (1.29)

7. Secondary Outcome: Change in Clinical Disease Activity Index (CDAI) From Baseline to Final Visit (Final Follow-up Visit)
Description: Clinical Disease Activity Index (CDAI) is the sum of 4 parameters: Swollen Joint Count 28 (SJC28, scored 0-28 with higher scores indicating higher disease activity) + Tender Joint Count 28 (TJC28, scored 0-28 with higher scores indicating higher disease activity) + Patient Global Assessment (PGA, scored on a visual analogue scale from 1-10 cm with higher scores indicating higher disease activity) + Physician Global Assessment (PhGA, scored on a visual analogue scale from 1-10 cm with higher scores indicating higher disease activity). CDAI scores range from 0 to 76 and indicate whether a participant is in remission or low, moderate or high activity; higher scores indicate higher disease activity. A negative change from baseline indicates improvement in condition.
  As this study was a non-interventional research initiative and no assessments/visits were mandated, the change in CDAI was only calculated for participants that had both baseline and final follow-up measurements.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: 56 participants were in the per protocol follow-up analysis set. Change in Clinical Disease Activity Index (CDAI) was calculated for participants who had both baseline and follow-up data required to calculate CDAI. For this measure, the mean change from baseline is based on 33 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 33
units on a scale | -5.59 (15.89)

8. Secondary Outcome: Change in Simple Disease Activity Index (SDAI) From Baseline to Final Visit (Final Follow-up Visit)
Description: Simple Disease Activity Index (SDAI) is the sum of the following 5 components to assess rheumatoid arthritis severity: Swollen Joint Count 28 (SJC28, scored 0-28 with higher scores indicating higher disease activity) + Tender Joint Count 28 (TJC28, scored 0-28 with higher scores indicating higher disease activity) + Patient Global Assessment (PGA, scored on a visual analogue scale from 1-10 cm with higher scores indicating higher disease activity) + Physician Global Assessment (PhGA, scored on a visual analogue scale from 1-10 cm with higher scores indicating higher disease activity) + C-reactive Protein (CRP). SDAI scores indicate whether a participant is in remission or low, moderate or high activity. A negative change in SDAI indicates improvement.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: 56 participants were in the per protocol follow-up analysis set. Change in Simple Disease Activity Index (SDAI) was calculated for participants who had both baseline and follow-up data required to calculate SDAI. For this measure, the mean change from baseline is based on 25 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 25
units on a scale | -6.28 (15.31)

9. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR) Response From Baseline to Final Visit (Final Follow-up Visit)
Description: European League Against Rheumatism (EULAR) response is based on change (improvement) in Disease Activity Score in 28 Joints score from baseline to last follow-up visit. DAS28 scores were broken into 3 categories: ≤3.2 at last follow-up (low disease activity), >3.2 and ≤ 5.1 at last follow-up (moderate or high disease activity), and DAS28 >5.1 at last follow-up (high disease activity). Then based on the category and magnitude of the change in DAS28 from baseline, the EULAR response of Good, Moderate or No Response was determined.
  DAS28 is an index for measuring disease activity in rheumatoid arthritis (RA). The index includes swollen joint counts (SJC) and tender joint counts (TJC), both scored 0-28 (higher scores indicate higher disease activity), as well as acute phase response determined as erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP), and patient global assessment (PGA) on a visual analogue scale (higher scores indicate higher disease activity).
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Measure: Number; unit: percentage of participants
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 56
percentage of participants
  Good response | 3.6
  Moderate response | 14.3
  No response | 28.6
  Missing | 44.6
  No follow-up visit/unable to calculate | 8.9

10. Secondary Outcome: Percentage of Participants With American College of Rheumatology 20% Improvement (ACR20) Response From Baseline to Final Visit (Final Follow-up Visit)
Description: American College of Rheumatology (ACR) 20, a patient must demonstrate a >= 20% improvement in tender and swollen joints (each scored 0-28 with higher scores indicating higher disease activity) as well as a 20% improvement in at least 3 of the following 5 parameters: patient global assessment (PGA, scored on a 1-10 scale with higher scores indicating higher disease activity), physician global assessment (PhGA, scored on a 1-10 scale with higher scores indicating higher disease activity), pain scale (scored on a 1-10 scale with higher scores indicating higher pain), functional questionnaire (scored on a 1-10 scale with higher scores indicating less function), and acute phase reactant (Erythrocyte Sedimentation Rate or C-reactive Protein).
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: 56 participants were in the per protocol follow-up analysis set. There were 27 participants with insufficient information to calculate ACR20 response and 5 participants have only baseline data. The percentages were calculated based on 56 participants.
Measure: Number; unit: percentage of participants
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 56
percentage of participants | 5.4

11. Secondary Outcome: Percentage of Participants With American College of Rheumatology 50% Improvement (ACR50) Response From Baseline to Final Visit (Final Follow-up Visit)
Description: American College of Rheumatology (ACR) 50, a patient must demonstrate a >= 50% improvement in tender and swollen joints (each scored 0-28 with higher scores indicating higher disease activity) as well as a 50% improvement in at least 3 of the following 5 parameters: patient global assessment (PGA, scored on a 1-10 scale with higher scores indicating higher disease activity), physician global assessment (PhGA, scored on a 1-10 scale with higher scores indicating higher disease activity), pain scale (scored on a 1-10 scale with higher scores indicating higher pain), functional questionnaire (scored on a 1-10 scale with higher scores indicating less function), and acute phase reactant (Erythrocyte Sedimentation Rate or C-reactive Protein).
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 56
percentage of participants | 1.8

12. Secondary Outcome: Percentage of Participants With American College of Rheumatology 70% Improvement (ACR70) Response From Baseline to Final Visit (Final Follow-up Visit)
Description: American College of Rheumatology (ACR) 70 a patient must demonstrate a >= 70% improvement in tender and swollen joints (each scored 0-28 with higher scores indicating higher disease activity) as well as a 70% improvement in at least 3 of the following 5 parameters: patient global assessment (PGA, scored on a 1-10 scale with higher scores indicating higher disease activity), physician global assessment (PhGA, scored on a 1-10 scale with higher scores indicating higher disease activity), pain scale (scored on a 1-10 scale with higher scores indicating higher pain), functional questionnaire (scored on a 1-10 scale with higher scores indicating less function), and acute phase reactant (Erythrocyte Sedimentation Rate or C-reactive Protein).
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: 56 participants were in the per protocol follow-up analysis set. There were 27 participants with insufficient information to calculate ACR70 response and 5 participants have only baseline data. The percentages were calculated based on 56 participants.
Measure: Number; unit: percentage of particpants
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 56
percentage of particpants | 1.8

13. Secondary Outcome: ACR-N From Baseline to Final Visit (Final Follow-up Visit)
Description: ACR-N is the index of improvement in rheumatoid arthritis, and is defined as the lowest of 3 values: percent change in the number of swollen joints (scored 0-28 with higher scores indicating higher disease activity), percent change in the number of tender joints (scored 0-28 with higher scores indicating higher disease activity), and the median of the other 5 measures in the American College of Rheumatology core data set-Patient's global assessment (PGA, scored on a 1-10 scale with higher scores indicating higher disease activity), physician's global assessment (PhGA, scored on a 1-10 scale with higher scores indicating higher disease activity), pain scale (scored on a 1-10scale with higher scores indicating higher pain), functional questionnaire (scored on a 1-10 scale with higher scores indicating less function), and acute phase reactant (Erythrocyte Sedimentation Rate or C-reactive Protein). Positive percent change indicates improvement. Negative percent change indicates worsening.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: 56 participants were in the per protocol follow-up analysis set. There were 27 participants with insufficient information to calculate ACR-N scores and 5 participants have only baseline data. ACR-N calculations were performed on data from 24 participants.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 24
percent change | -15.4 (43.6)

14. Secondary Outcome: Change in Routine Assessment of Patient Index Data (RAPID3) From Baseline to Final Visit (Final Follow-up Visit)
Description: Routine Assessment of Patient Index Data (RAPID3) was calculated by summing three measures: physical function (0 to 10 with higher scores indicating less function), pain (0 to 10 with higher scores indicating higher pain), and patient global assessment (0 to 10 with higher scores indicating the participant was doing very poorly considering the ways in which the illness was affecting them). As this study was a non-interventional research initiative and no assessments or visits were mandated, the change in RAPID3 was only calculated for participants that had measurements at both baseline and final follow-up.
  RAPID3 scores range from 0 to 30 with higher scores meaning worse condition. A negative change from baseline indicates improvement in condition.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: 56 participants were in the per protocol follow-up analysis set. Change in Routine Assessment of Patient Index Data (RAPID3) was calculated for participants who had both baseline and follow-up data required to calculate RAPID3. For this measure, the mean change from baseline is based on 33 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 33
units on a scale | -2.06 (5.45)

15. Secondary Outcome: Change in Multidimensional Health Assessment Questionnaire (MDHAQ) Function (FN) Component From Baseline to Final Visit (Final Follow-up Visit)
Description: The change in Multidimensional Health Assessment Questionnaire (MDHAQ) - function (FN) was assessed by asking participants to score the performance of multiple activities as "without any difficulty" (score of 0), "with some difficulty" (score of 1), "with much difficulty" (score of 2) or "unable to do" (score of 3). The results were summed and divided by 3 to give a score from 0 to10. A negative change from baseline indicates improvement. As this study was a non-interventional research initiative and no assessments or visits were mandated, the change in function was only calculated for participants that had measurements at both baseline and final follow-up.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: 56 participants were in the per protocol follow-up analysis set. Change in Multidimensional Health Assessment Questionnaire (MDHAQ) - Function (FN) was calculated for participants who had both baseline and follow-up FN data. For this measure, the mean change from baseline is based on 33 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 33
units on a scale | -0.05 (1.66)

16. Secondary Outcome: Change in Multidimensional Health Assessment Questionnaire (MDHAQ) Psychological Status (PS) Component From Baseline to Final Visit (Final Follow-up Visit)
Description: The change in Multidimensional Health Assessment Questionnaire (MDHAQ) - Psychological status (PS) was assessed by asking participants to score how they were sleeping, dealing with anxiety/nervousness, and dealing with depression as "without any difficulty" (score of 0), "with some difficulty" (score of 1.1), "with much difficulty" (score of 2.2) or "unable to do" (score of 3.3). The results were summed to give a score ranging from 0 to 9.9. A negative change from baseline indicates improvement. As this study was a non-interventional research initiative and no assessments or visits were mandated, the change in psychological status was only calculated for participants that had measurements at both baseline and final follow-up.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: 56 participants were in the per protocol follow-up analysis set. Change in Multidimensional Health Assessment Questionnaire (MDHAQ) - Psychological status (PS) was calculated for participants who had both baseline and follow-up PS data. For this measure, the mean change from baseline is based on 33 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 33
units on a scale | 0.17 (2.45)

17. Secondary Outcome: Change in Multidimensional Health Assessment Questionnaire (MDHAQ) Pain (PN) Component From Baseline to Final Visit (Final Follow-up Visit)
Description: Multidimensional Health Assessment Questionnaire (MDHAQ) - pain (PN) scoring was gathered using a 0-10 scale where 0 corresponded to "No Pain" and 10 to "Pain as bad as it could be" because of the condition (over the past week). A negative change from baseline indicates improvement. As this study was a non-interventional research initiative and no assessments or visits were mandated, the change in pain was only calculated for participants that had measurements at both baseline and final follow-up.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: 56 participants were in the per protocol follow-up analysis set. Change in Multidimensional Health Assessment Questionnaire (MDHAQ) - Pain (PN) was calculated for participants who had both baseline and follow-up PN data. For this measure, the mean change from baseline is based on 33 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 33
units on a scale | -0.62 (2.44)

18. Secondary Outcome: Change in Multidimensional Health Assessment Questionnaire (MDHAQ) the Rheumatoid Arthritis Disease Activity Index (RADAI) Patient Self-report Joint Count (PTJT) Component From Baseline to Final Visit (Final Follow-up Visit)
Description: For the Change in Multidimensional Health Assessment Questionnaire (MDHAQ) - the Rheumatoid Arthritis disease Activity Index (RADAI) patient self-report joint count (PTJT), participants were asked to score the amount of pain they were experiencing in each of 16 joints (left joint, left wrist, right shoulder etc.) as "None" (score of 0), "Mild" (score of 1), "Moderate" (score of 2) or "Severe" (score of 3). The raw 0-48 score is adjusted to 0-10 using a scoring template. A negative change from baseline indicates improvement. As this study was a non-interventional research initiative and no assessments or visits were mandated, the change in PTJT was only calculated for participants that had measurements at both baseline and final follow-up.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: 56 participants were in the per protocol follow-up analysis set. Change in Multidimensional Health Assessment Questionnaire (MDHAQ) - RADAI patient self-report joint count (PTJT) was calculated for participants who had both baseline and follow-up data. For this measure, the mean change from baseline is based on 33 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 33
units on a scale | -0.29 (2.04)

19. Secondary Outcome: Change in Multidimensional Health Assessment Questionnaire (MDHAQ) Neck and Back (NB) Component From Baseline to Final Visit (Final Follow-up Visit)
Description: For the Multidimensional Health Assessment Questionnaire (MDHAQ) - neck and back (NB), participants were asked to score the amount of pain they were experiencing in their neck and back as "None" (score of 0), "Mild" (score of 1), "Moderate" (score of 2) or "Severe" (score of 3). The raw 0-6 score was adjusted to 0-10. A negative change from baseline indicates improvement. As this study was a non-interventional research initiative and no assessments or visits were mandated, the change in NB measure was only calculated for participants that had measurements at both baseline and final follow-up.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: 56 participants were in the per protocol follow-up analysis set. Change in Multidimensional Health Assessment Questionnaire (MDHAQ) - neck and back (NB) was calculated for participants who had both baseline and follow-up NB data. For this measure, the mean change from baseline is based on 33 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 33
units on a scale | -0.35 (2.75)

20. Secondary Outcome: Change in Multidimensional Health Assessment Questionnaire (MDHAQ) Patient Global Assessment (PTGL) Component From Baseline to Final Visit (Final Follow-up Visit)
Description: Multidimensional Health Assessment Questionnaire (MDHAQ) - patient global assessment (PTGL) was measured by asking the participant to rate on a 0 to 10 scale how they were doing considering all of the ways in which their illness and health conditions affected them: 0 - Very Well, 10 - Very Poor. A negative change from baseline indicates improvement. As this study was a non-interventional research initiative and no assessments or visits were mandated, the change in PTGL was only calculated for participants that had measurements at both baseline and final follow-up.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: 56 participants were in the per protocol follow-up analysis set. Change in Multidimensional Health Assessment Questionnaire (MDHAQ) - patient global assessment (PTGL) was calculated for participants who had both baseline and follow-up PTGL data. For this measure, the mean change from baseline is based on 33 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 33
units on a scale | -0.53 (2.91)

21. Secondary Outcome: Change in Multidimensional Health Assessment Questionnaire (MDHAQ) Review of Symptoms (ROS) Component From Baseline to Final Visit (Final Follow-up Visit)
Description: Multidimensional Health Assessment Questionnaire (MDHAQ) - review of symptoms (ROS) was gathered using a symptom checklist and was calculated by summing the total number of items checked (0 to 60 symptoms could be checked). A negative change from baseline indicates improvement. As this study was a non-interventional research initiative and no assessments or visits were mandated, the change in MDHAQ ROS was only calculated for participants that had measurements at both baseline and final follow-up.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: 56 participants were in the per protocol follow-up analysis set. Change in Multidimensional Health Assessment Questionnaire (MDHAQ) - review of symptoms (ROS) was calculated for participants who had both baseline and follow-up ROS data. For this measure, the mean change from baseline is based on 33 participants.
Measure: Mean (Standard Deviation); unit: number of symptoms
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 33
number of symptoms | -0.3 (5.2)

22. Secondary Outcome: Change in Multidimensional Health Assessment Questionnaire (MDHAQ) Morning Stiffness Component From Baseline to Final Visit (Final Follow-up Visit)
Description: The duration of morning stiffness was the amount of time participants experienced stiffness after waking up in the morning (over the last week). This measure was collected at baseline and at the last follow-up visit. A negative change from baseline indicates improvement. As this study was a non-interventional research initiative and no assessments or visits were mandated, the change in duration of morning stiffness was only calculated for participants that had measurements at both baseline and final follow-up.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: 56 participants were in the per protocol follow-up analysis set. Change in Multidimensional Health Assessment Questionnaire (MDHAQ) - morning stiffness, minutes (past week) was calculated for participants who had both baseline and follow-up data. For this measure, the mean change from baseline is based on 30 participants.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 30
minutes | -2.5 (67.0)

23. Secondary Outcome: Change in Multidimensional Health Assessment Questionnaire (MDHAQ) "How do You Feel Today (Compared to One Week Ago)" Component From Baseline to Final Visit (Final Follow-up Visit)
Description: The Multidimensional Health Assessment Questionnaire (MDHAQ) - how do you feel today compared to one week ago question was scored as follows: 1: Much Better, 2: Better, 3: The Same, 4: Worse, 5: Much Worse. A negative change from baseline indicates improvement. As this study was a non-interventional research initiative and no assessments or visits were mandated, the change in "How do you feel" measure was only calculated for participants that had measurements at both baseline and final follow-up.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: 56 participants were in the per protocol follow-up analysis set. Change in Multidimensional Health Assessment Questionnaire - How do you feel today (compared to 1wk ago) from Baseline to Final Visit was calculated for participants who had both baseline and follow-up data. For this measure, the mean change from baseline is based on 33 participants.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 33
units on a scale | -0.2 (0.8)

24. Secondary Outcome: Change in Multidimensional Health Assessment Questionnaire (MDHAQ) Exercise (EX) Component From Baseline to Final Visit (Final Follow-up Visit)
Description: The exercise aerobically for at least one-half hour (30 minutes) measure of the multidimensional health assessment questionnaire (MDHAQ) was scored as follows: "3 or more times a week" (3), "1-2 times per week" (2), "1-2 times per month" (1), "Do not exercise regularly" (0), "Cannot exercise due to disability/handicap" (-1). As this study was a non-interventional research initiative and no assessments or visits were mandated, the change in MDHAQ exercise measure was only calculated for participants that had measurements at both baseline and final follow-up.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: 56 participants were in the per protocol follow-up analysis set. Change in Multidimensional Health Assessment Questionnaire (MDHAQ) - exercise (EX) was calculated for participants who had both baseline and follow-up EX data. For this measure, the mean change from baseline is based on 33 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 33
units on a scale | -0.1 (1.1)

25. Secondary Outcome: Change in Multidimensional Health Assessment Questionnaire (MDHAQ) Fatigue (FAT) Component From Baseline to Final Visit (Final Follow-up Visit)
Description: Multidimensional Health Assessment Questionnaire (MDHAQ) - fatigue (FAT) scoring was gathered using a 0-10 scale where 0 corresponded to "Fatigue is no problem" and 10 to "Fatigue is a major problem" over the past week. A negative change from baseline indicates improvement. As this study was a non-interventional research initiative and no assessments or visits were mandated, the change in fatigue was only calculated for participants that had measurements at both baseline and final follow-up.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: 56 participants were in the per protocol follow-up analysis set. Change in Multidimensional Health Assessment Questionnaire (MDHAQ) - fatigue (FAT) was calculated for participants who had both baseline and follow-up FAT data. For this measure, the mean change from baseline is based on 33 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 33
units on a scale | -0.12 (3.14)

26. Secondary Outcome: Change in Multidimensional Health Assessment Questionnaire (MDHAQ) Recent Medical History Component From Baseline to Final Visit (Final Follow-up Visit)
Description: Multidimensional Health Assessment Questionnaire (MDHAQ) - recent medical history was gathered using a medical history checklist and was calculated by summing the total number of items checked "Yes" (0 to 12 items could be checked). A negative change from baseline indicates fewer items were checked at the follow-up visit. As this study was a non-interventional research initiative and no assessments or visits were mandated, the change in MDHAQ recent medical history was only calculated for participants that had measurements at both baseline and final follow-up.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: 56 participants were in the per protocol follow-up analysis set. Change in Multidimensional Health Assessment Questionnaire (MDHAQ) - recent medical history was calculated for participants who had both baseline and follow-up recent medical history data. For this measure, the mean change from baseline is based on 33 participants.
Measure: Mean (Standard Deviation); unit: number of items checked
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 33
number of items checked | -0.2 (1.2)

27. Secondary Outcome: Corticosteroid Sparing Effect - Change in Total Daily Prednisone Dose From Baseline to Final Visit (Final Follow-up Visit)
Description: The change in total daily prednisone from baseline to follow-up (whether the patient was taking RAYOS or returned to conventional prednisone) was calculated for all participants.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 56
milligrams | -0.96 (3.61)

28. Secondary Outcome: Assessment of Unsolicited Adverse Events
Description: Please refer to the safety section for further details.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 75
Participants | 11

29. Secondary Outcome: Assessment of Unsolicited Serious Adverse Events
Description: Please refer to the safety section for further details.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 75
Participants | 1

30. Other Pre Specified Outcome: Correlation Between Vectra DA and DAS28 at Each Assessed Time Point
Description: Vectra DA and DAS28 data were collected, however not analyzed or correlated.
Time Frame: Baseline to Last Follow up visit (up to 18.7 weeks)
Population: Analysis and correlations were not completed for this outcome measure.
Arm/Group | Delayed-release Prednisone (RAYOS)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From signing of informed consent form through the last follow-up visit (up to 18.7 weeks)
Arm/Group | Delayed-release Prednisone (RAYOS)
Serious Adverse Events (participants affected / at risk) | 1/75
Other Adverse Events (participants affected / at risk) | 11/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Delayed-release Prednisone (RAYOS) (N=75)
Abdominal Pain (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Delayed-release Prednisone (RAYOS) (N=75)
High Blood Pressure (Cardiac disorders) | 1
Abdominal Pain/Nausea (Gastrointestinal disorders) | 1
Insomnia (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Animal Bite (Injury, poisoning and procedural complications) | 1
Worsening of Joint Pain (Musculoskeletal and connective tissue disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Ankle Pain (Musculoskeletal and connective tissue disorders) | 1
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1
Elevated blood glucose (Metabolism and nutrition disorders) | 1
General malaise leading to loss of appetite (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Physician agrees to obtain written consent of Horizon prior to publishing or presenting any results of the SUNRAY Observational Study.